CLINICAL TRIAL: NCT04410289
Title: A Prospective Randomized Pilot Study to Define and Validate the Standard 'Sniffing Position' in Infants and Toddlers.
Brief Title: Defining the 'Sniffing Position" in Infants and Toddlers - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13188
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Airway Management; Infant ALL; Children, Only; Endotracheal Intubation
Keywords: pediatric intubation; direct laryngoscopy; sniffing position; external auditory meatus; pediatric anesthesia; pediatric airway management
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After induction of general anesthesia, and prior to direct laryngoscopy, patients in the intervention group were positioned using props horizontally aligning the external auditory meatus (EAM) with the sternal notch (SN) and the chin with the sinciput. A lateral side-profile photograph was taken for latter analysis and an Intubation Difficulty Scale (IDS) score card completed.
  Interventions: Procedure: Airway positioning per specified protocol followed by Direct Laryngoscopy and Endotracheal Intubation
- Control Group (Active Comparator): After induction of general anesthesia, and prior to direct laryngoscopy, patients in the control group were positioned freely according to the provider's preference. A lateral side-profile photograph was taken for latter analysis and an Intubation Difficulty Scale (IDS) score card completed.
  Interventions: Procedure: Airway positioning per provider preference followed by Direct Laryngoscopy and Endotracheal Intubation

INTERVENTIONS:
Procedure: Airway positioning per specified protocol followed by Direct Laryngoscopy and Endotracheal Intubation — Positioning of the patient's head and neck for the purpose of direct laryngoscopy and endotracheal intubation
  Arms: Intervention Group
Procedure: Airway positioning per provider preference followed by Direct Laryngoscopy and Endotracheal Intubation — Positioning of the patient's head and neck for the purpose of direct laryngoscopy and endotracheal intubation
  Arms: Control Group

SUMMARY:
The "sniffing position" is widely accepted as a favorable position for direct laryngoscopy (DL) in both pediatric and adult patients. External anatomical markers are well documented to confirm proper 'sniffing position' in adults, but data on their use in the pediatric population is sparse. The investigators propose to define these markers in young children and investigate whether patients positioned using this standardized approach have better intubating conditions than those positioned randomly per the preference of the anesthesiologist.

DETAILED DESCRIPTION:
The procedure of endotracheal intubation in adults and children is a continuum, and begins with proper head positioning prior to direct laryngoscopy (DL). It is an accepted paradigm that proper positioning optimizes intubating conditions, and decreases subsequent airway maneuvers and manipulation.

The sniffing position is an accepted airway positioning concept in pediatric airway management, and continues to be recommended by experts and textbooks in the field. Anatomical peculiarities such as the large head relative to the torso in infants and toddlers is assumed to put the head in proper position when gently extended. However, reproducible parameters to confirm optimal head positioning remain vague and unclear. In the absence of objective and measurable markers, practitioners position infants and toddlers according to their individual preferences, and as such the procedure lacks definition and objective clarity.

The investigators plan to recruit 40 healthy patients between the ages of 1 month - 48 months and randomize them to be positioned either according to a predetermined algorithm or positioned freely according to the provider's preference. Patients randomized to the intervention group will be positioned with the aim to horizontally align the external auditory meatus (EAM) with the sternal notch (SN).

In summary, the study aims to define the sniffing position for infants and toddlers using reproducible objective secondary markers, and investigate whether a systematic approach to positioning using such markers improves direct laryngoscopic outcomes in the young pediatric patient population.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants and toddlers undergoing non-emergent surgery under general anesthesia with an oral endotracheal tube

Exclusion Criteria:

* neonates (infants under 1 month of age), infants and toddlers with congenital syndromes affecting the airway, and patients undergoing emergency surgery.

Ages: 1 Month to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Difference in Intubation Difficulty Scale (IDS) Score | The brief time involved (5-10 minutes) involving the process of head positioning, direct laryngoscopy and endotracheal intubation.
  To assess the difference in IDS scores between the study and control groups

SECONDARY OUTCOMES:
Angles of Deviation of the EAM-SN plane and Chin-Sinciput Plane from the Horizontal | Post-hoc analysis using a computer program to calculate angles. 10 minutes per patient.
  Secondary outcome was to analyze and compare the degree of alignment or nonalignment of the EAM-SN plane and the sinciput-chin plane in both groups. Angles of deviation of the EAM-SN and chin-sinciput plane were measured in each cohort based on photographic data collected. A positive angle deviation indicated head flexion and a negative angle indicated head extension.

CONTACTS AND LOCATIONS:
Overall Officials: Aman Kalra, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akihisa Y, Hoshijima H, Maruyama K, Koyama Y, Andoh T. Effects of sniffing position for tracheal intubation: a meta-analysis of randomized controlled trials. Am J Emerg Med. 2015 Nov;33(11):1606-11. doi: 10.1016/j.ajem.2015.06.049. Epub 2015 Jun 23. PMID 26227445
- [Background] El-Orbany M, Woehlck H, Salem MR. Head and neck position for direct laryngoscopy. Anesth Analg. 2011 Jul;113(1):103-9. doi: 10.1213/ANE.0b013e31821c7e9c. Epub 2011 May 19. PMID 21596871
- [Background] Greenland KB, Eley V, Edwards MJ, Allen P, Irwin MG. The origins of the sniffing position and the Three Axes Alignment Theory for direct laryngoscopy. Anaesth Intensive Care. 2008 Jul;36 Suppl 1:23-7. doi: 10.1177/0310057X0803601s05. PMID 18724555
- [Background] Greenland KB, Edwards MJ, Hutton NJ. External auditory meatus-sternal notch relationship in adults in the sniffing position: a magnetic resonance imaging study. Br J Anaesth. 2010 Feb;104(2):268-9. doi: 10.1093/bja/aep390. No abstract available. PMID 20086071
- [Background] Prakash S, Rapsang AG, Mahajan S, Bhattacharjee S, Singh R, Gogia AR. Comparative evaluation of the sniffing position with simple head extension for laryngoscopic view and intubation difficulty in adults undergoing elective surgery. Anesthesiol Res Pract. 2011;2011:297913. doi: 10.1155/2011/297913. Epub 2011 Oct 29. PMID 22110497
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Horton WA, Fahy L, Charters P. Defining a standard intubating position using "angle finder". Br J Anaesth. 1989 Jan;62(1):6-12. doi: 10.1093/bja/62.1.6. PMID 2917111
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Kim BR, Kim HS. Effect of head position on laryngeal visualisation with the McGrath MAC videolaryngoscope in paediatric patients: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):528-34. doi: 10.1097/EJA.0000000000000448. PMID 26986776
- [Background] Vialet R, Nau A, Chaumoitre K, Martin C. Effects of head posture on the oral, pharyngeal and laryngeal axis alignment in infants and young children by magnetic resonance imaging. Paediatr Anaesth. 2008 Jun;18(6):525-31. doi: 10.1111/j.1460-9592.2008.02530.x. Epub 2008 Mar 18. PMID 18363622
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Greenland KB, Edwards MJ, Hutton NJ, Challis VJ, Irwin MG, Sleigh JW. Changes in airway configuration with different head and neck positions using magnetic resonance imaging of normal airways: a new concept with possible clinical applications. Br J Anaesth. 2010 Nov;105(5):683-90. doi: 10.1093/bja/aeq239. Epub 2010 Sep 15. PMID 20846964